CLINICAL TRIAL: NCT01301521
Title: Cinnamon Trial-Assessment of the effeCt of lIfestyle iNtervention Plus Water-soluble ciNnAMon Extract On loweriNg Blood Glucose in Pre-diabetics: A Randomized, Double-blind, Multicenter, Placebo Controlled TRIAL.
Brief Title: Cinnamon Trial-lIfestyle iNtervention Plus Water-soluble Cinnamon Extract On loweriNg Blood Glucose in Pre-diabetics
Acronym: Cinnamon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FWH20110035H
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Diabetes; Pre-Diabetes
Keywords: Pre-Diabetes; cinnamon
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance | interventions — cinnulin PF

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinnulin PF (Experimental): Will take (by mouth) 2 gelatin capsules that contains 1 gram (2-500 mg capsules) water-soluble cinnamon extract (Cinnulin PF) once a day for 1 year plus 1 year of follow-up plus standard of care aggressive lifestyle therapy.
  Interventions: Drug: water-soluble cinnamon extract (Cinnulin PF)
- Placebo (Placebo Comparator): Will take (by mouth) 2 placebo capsules (gelatin capsule filled with wheat bran) once a day for 1 year plus 1 year of follow-up plus standard of care aggressive lifestyle therapy.
  Interventions: Drug: water-soluble cinnamon extract (Cinnulin PF)

INTERVENTIONS:
Drug: water-soluble cinnamon extract (Cinnulin PF) — Will take (by mouth) 1 gelatin capsule that contains 1 gram water-soluble cinnamon extract (Cinnulin PF) once a day for 12 months plus standard of care aggressive lifestyle therapy
  Other Names: Cinnulin PF

SUMMARY:
The purpose of this study is to assess whether water-soluble cinnamon extract plus aggressive lifestyle intervention is effective in lowering blood glucose in pre-diabetic patients when compared to aggressive lifestyle therapy plus placebo.

DETAILED DESCRIPTION:
We are studying whether water-soluble cinnamon extract (Cinnulin PF) plus standard of care aggressive lifestyle therapy is effective in lowering blood glucose when compared to placebo plus standard of care aggressive life style therapy. Eligible subjects will be recruited from any form and any stage of "standard" lifestyle intervention for pre-diabetes at an individual base. "Standard" lifestyle intervention for pre-diabetes could include Group Lifestyle Balance (GLB), nutrition classes, Better Body/Better Life, or anything an investigator certifies as standard practice at that base. Subjects will take either 1 gram (2-500 milligram (mg) capsules) of water-soluble cinnamon extract (Cinnulin PF) or 2 placebo pills (gelatin capsule filled with wheat bran) once a day for 1 year plus 1 additional year of follow-up. This is a randomized, double-blind, multicenter, placebo-controlled study which will enroll subjects at the Mike O'Callaghan Federal Medical Center (MOFMC), Wilford Hall Ambulatory Surgical Center (WHASC), David Grant Medical Center (DGMC), Eglin Air Force Base (Eglin), and Offutt Air Force Base (Offutt). All subjects will be MOFMC, WHASC, DGMC, Eglin, and Offutt DoD beneficiaries. Informed Consent and HIPAA Authorization will be obtained. After randomization, subjects will receive either 1 gram (2-500 mg capsules) of water-soluble cinnamon extract or placebo from the pharmacy--thus investigators and subjects will be blinded as to if they are taking Cinnulin PF or 2 placebo pills. Subjects will be permitted to have usual medical care for other co-morbid, preventive, and acute conditions. Analysis will be performed using intention-to-treat principles for missing data (the carry-forward method to impute missing data will be used). Subjects will bring in any remaining water-soluble cinnamon extract or placebo to determine adherence rates to the study protocol.

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

Patients will be MOFMC, WHASC, DGMC, Eglin, and Offutt DoD beneficiaries, ages 18-65 years.

Diagnosis of pre-diabetes (defined as a fasting plasma glucose (FPG) 100-125mg/dl, Hemoglobin A1c 5.7-6.4%, or a 2-hour oral glucose tolerance test (OGTT) 140-199).

Exclusion:

Patients who are less than 18 yrs of age or greater than 65 years of age.

Patients who are known to have or develop during the study any of the following upon review of their medical record:

* Diabetes Mellitus (defined as fasting plasma glucose (FPG) greater than 126mg/dl, hemoglobin A1C greater than 6.5%, or a 2-hour oral glucose tolerance test (OGTT) greater than 200mg/dl)
* Stage 3 kidney disease or worse
* Renal insufficiency defined as a glomerular filtration rate (gfr) of less than 60ml
* Celiac disease
* Insulinoma
* Cushing's disease
* Hyperthyroidism
* Acromegaly
* Pheochromocytoma
* Addison's disease
* Galactosemia
* Glycogen storage disease
* Hereditary fructose intolerance

Patients taking any of the following:

* Cinnamon as a dietary supplement
* Daily oral steroids
* Warfarin
* Hypoglycemic medication
* Weight loss medication
* Digoxin, lithium, phenytoin, & theophylline (due to their narrow therapeutic indices) Patients who are pregnant or breast feeding Patients with a known allergy to cinnamon Patients with a known allergy to wheat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, M.D., Principal Investigator — Mike O'Callaghan Federal Hospital/Nellis Air Force Base
Locations (4):
- United States (4):
  - Travis Air Force Base, Travis Air Force Base, California
  - Eglin Air Foce Base, Eglin Air Force Base, Florida
  - Offutt Air Force Base, Offutt Air Force Base, Nebraska
  - Wilford Hall Ambulatory Surgical Center, Lackland Air Force Base, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crawford P, Thai C, Obholz J, Schievenin J, True M, Shah SA, Hallgren J, Clark J, Sharon D. Assessment of the effeCt of lIfestyle iNtervention plus water-soluble ciNnAMon extract On loweriNg blood glucose in pre-diabetics, a randomized, double-blind, multicenter, placebo controlled trial: study protocol for a randomized controlled trial. Trials. 2016 Jan 5;17:9. doi: 10.1186/s13063-015-1138-7. PMID 26732017

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cinnulin PF | Placebo
Started | 116 | 113
Completed | 47 | 43
Not Completed | 69 | 70

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinnulin PF | Placebo | Total
Number analyzed (Participants) | 116 | 113 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 116 | 113 | 229
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 125
  Male | 52 | 52 | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 9 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 6 | 7
  Black or African American | 38 | 20 | 58
  White | 53 | 69 | 122
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Water-soluble Cinnamon
Description: Does water-soluble cinnamon extract delay the onset of diabetes or extend the time to diagnosis of diabetes in pre-diabetic patients who are already undergoing aggressive lifestyle therapy?
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cinnulin PF | Placebo
Number analyzed (Participants) | 47 | 43
Participants
  diabetes conversion: yes | 15 | 11
  diabetes conversion: no | 32 | 32

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cinnulin PF | Placebo
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/113
Other Adverse Events (participants affected / at risk) | 41/116 | 30/113
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cinnulin PF (N=116) | Placebo (N=113)
Unrelated to Medicine (General disorders) | 27 (27) | 28 (28)
Medication Reaction (General disorders) | 14 (14) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT01301521/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT01301521/ICF_001.pdf